CLINICAL TRIAL: NCT03697850
Title: Phase II Study of Maintenance Anti-PD-L1 Treatment With Atezolizumab After Chemo-radiotherapy for Muscle-infiltrating Bladder Cancer Patients Not Eligible for Radical Cystectomy: Bladder Sparing
Brief Title: Atezolizumab After Chemo-radiotherapy for MIBC Patients Not Eligible for Radical Cystectomy
Acronym: BladderSpar
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UC-0160/1715; 2018-001807-35 (EudraCT Number)
Record Dates: First submitted 2018-10-02; First posted 2018-10-05 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2024-12

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- atezolizumab (Experimental): Anti-PD-L1 immunotherapy: atezolizumab (1200 mg) administered IV over 1 h every 3 weeks for 12 months (18 injections). Beginning 30 days (±5 days) after chemo-radiotherapy.
  Interventions: Drug: Atezolizumab

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab after adjuvant radio-chemotherapy for the treatment of patients with muscle-invasive bladder cancer not eligible for radical cystectomy

SUMMARY:
Patients older than ≥18 years, with muscle-invasive bladder cancer unfit for radical cystectomy because of age, comorbidities, and/or patient's refusal.

This study is designed as a multicentre, single-arm phase II study.

ELIGIBILITY:
Selection phase

Inclusion Criteria:

1. Muscle-invasive bladder cancer (MIBC) pT2-T3 histologically confirmed:

   Urothelial and squamous cell histological types are allowed. De novo MIBC or after a history of non-muscle-invasive bladder cancer.
2. Complete transurethral resection of bladder tumour (TURBT), either:

   within 6 weeks of selection if no chemotherapy was administered, or before starting chemotherapy.
3. Patients for which chemo-radiotherapy is planned
4. No major pelvic involvement: pelvic nodes ≤15 mm on CT scan.
5. No distant metastasis.
6. Patient unfit for radical cystectomy because of age, comorbidities, or patient's refusal.
7. Patients ≥18 years old
8. Eastern Cooperative Oncology Group (ECOG) performance status ≤2.
9. Life expectancy ≥12 months.
10. Haematological and biological parameters:

    White blood cell count ≥4000/mm³ Platelet count ≥100000 cells/mm³ Haemoglobin level ≥9 g/dL or corrected after transfusion Adequate renal function: clearance >50 mL/min (Cockcroft). Adequate hepatic function: Aspartate aminotransferase (AST [SGOT]) and Alanine aminotransferase (ALT [SGPT]) ≤2.5 x upper limit of normal (ULN), or ≤3.5 x ULN in the case of concurrent disease with known etiology and for which a corrective treatment is possible.
11. Patients of childbearing potential who agree to use a medically acceptable method of contraception during the study and for 120 days after the last study treatment. Women must have a negative urine or serum pregnancy test before receiving the study treatment and within 14 days prior to selection.
12. Patients having provided written informed consent prior to any study-related procedures.
13. Patients affiliated to the social security scheme.
14. Patients willing and able to comply with the scheduled visits, treatment plan, laboratory tests, and other study procedures indicated in the protocol.
15. Patient consents to the use of their collected tumour specimen, as well as, blood samples as detailed in the protocol for future scientific research which includes but not limited to DNA, RNA, and protein-based biomarker detection.

Exclusion Criteria:

1. Prior pelvic irradiation.
2. MIBC histology other than urothelial or squamous cell carcinomas (e.g., adenocarcinomas, micropapillary, sarcomas, or small cell histological types).
3. History of neoplastic disease, during the 3 years before selection, except completely resected cutaneous basal-cell carcinomas, carcinoma in-situ or localised prostate cancer without biochemical recurrence following definitive treatment.
4. Prior treatment with CD137 agonists or immune checkpoint inhibitors, including anti-cytotoxic T lymphocyte-associated antigen 4 (anti-CTLA-4), anti-programmed death-1 receptor (anti-PD-1), and anti-programmed death-ligand 1 (anti-PD-L1) therapeutic antibodies.
5. Contraindications for pelvic radiotherapy (e.g., inflammatory bowel disease).
6. History of immunodeficiency, including HIV infection, or systemic steroid therapy for any other disease.
7. A history of active autoimmune disease, except autoimmune-related hypothyroidism and type I diabetes mellitus (see appendix 5).
8. History of severe allergic anaphylactic reactions to chimeric, human or humanised antibodies, or fusion proteins.
9. Known hypersensitivity to Chinese hamster ovary (CHO) cell products or any component of the atezolizumab formulation.
10. Prior allogeneic stem cell or solid organ transplant.
11. Patients with the following severe acute co-morbidity are not eligible:

    Unstable angina or congestive heart failure that required hospitalisation in the 6 months before selection.

    Transmural myocardial infarction in the 6 months prior to selection. Acute bacterial or fungal infection requiring intravenous antibiotics at selection.

    Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalisation or precluding study therapy at the time of selection.

    Severe hepatic disease: Child-Pugh Class B or C.
12. Patients with any other disease or illness which requires hospitalisation or is incompatible with the study treatment are not eligible.
13. Patients unable to comply with study obligations for geographic, social, or physical reasons, or who are unable to understand the purpose and procedures of the study.
14. Patients enrolled in another therapeutic study within 30 days of selection.
15. Pregnant or breast feeding women.
16. Person deprived of their liberty or under protective custody or guardianship.

Inclusion phase

Inclusion Criteria:

1. Patients who have received standard (chemo)-radiotherapy ≥60 gray (Gy) or equivalent on the bladder according to the local practice.
2. The first administration of atezolizumab must be performed 30 (+/-5) days after the last session of radiotherapy (RT).
3. ECOG performance status ≤2.
4. Haematological and biological parameters:

   White blood cell count ≥3000/mm³ Platelet count ≥100000 cells/mm³ Haemoglobin level ≥9 g/dL or corrected after transfusion Adequate renal function: clearance >50 mL/min (Cockcroft) Adequate hepatic function: AST (SGOT) and ALT (SGPT) ≤2.5 x ULN, or ≤3.5 x ULN in the case of concurrent disease with known etiology and for which a corrective treatment is possible.
5. Patients of childbearing potential who agree to use a medically acceptable method of contraception during the study and for 120 days after the last study treatment. Women must have a negative urine or serum pregnancy test before receiving the study treatment and within 14 days prior to inclusion.
6. Patients having provided written informed consent prior to any study-related procedures.
7. Patients willing and able to comply with the scheduled visits, treatment plan, laboratory tests, and other study procedures indicated in the protocol.
8. Patient consents to the use of their collected tumour specimen, as well as, blood samples as detailed in the protocol for future scientific research which includes but not limited to DNA, RNA, and protein-based biomarker detection.

Exclusion Criteria:

The same non-inclusion criteria of the selection phase have to be respected.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2018-12-14 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2029-02-15 (Estimated)

PRIMARY OUTCOMES:
Disease Free Survival | 2 years
  Disease Free Survival is defined as the delay between date of inclusion and tumour relapse (local, regional, or distant) or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Local control rate | 2 years
  Local control rate will be evaluated by cystoscopy. The presence of non-muscle-invasive or muscle-invasive bladder cancers will be considered as a local failure. To be defined as locally controlled, the bladder must be completely free of tumour.
Local control rate | 5 years
  Local control rate will be evaluated by cystoscopy. The presence of non-muscle-invasive or muscle-invasive bladder cancers will be considered as a local failure. To be defined as locally controlled, the bladder must be completely free of tumour.
Disease Free Survival | 5 years
  Disease Free Survival is defined as the delay between date of inclusion and tumour relapse (local, regional, or distant) or death from any cause, whichever occurs first.
Overall Survival | 2 years
  Overall Survival is defined as the delay between the date of inclusion and the date of death, from any cause.
Overall Survival | 5 years
  Overall Survival is defined as the delay between the date of inclusion and the date of death, from any cause.
Incidence of Treatment-Emergent Adverse Events | 2 years
  The tolerance and safety will be evaluated by toxicity (acute [<6 months after the start of atezolizumab] and late [≥6 months after the start of atezolizumab]), assessed using the NCI CTCAE v5.0
Incidence of Treatment-Emergent Adverse Events | 5 years
  The tolerance and safety will be evaluated by toxicity (acute [<6 months after the start of atezolizumab] and late [≥6 months after the start of atezolizumab]), assessed using the NCI CTCAE v5.0
Quality of Life Core Questionnaire - Cancer Patients (QLQ-C30) | 5 years
  Quality of life
Quality of Life Core Questionnaire - Bladder Cancer Muscle Invasive (QLQ-BLM30) | 5 years
  Quality of Life
Quality of Life Core Questionnaire - Elderly Cancer Patients (QLQ-ELD14) | 5 years
  Quality of Life
G8 oncodage | 5 years
  Quality of Life

CONTACTS AND LOCATIONS:
Overall Officials: Christophe HENNEQUIN, Prof, Principal Investigator — Hôpital Saint Louis
Locations (12):
- France (12):
  - Institut Bergonie, Bordeaux
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Georges Francois Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Icm Val D'Aurelle, Montpellier
  - Centre Azureen de Cancerologie, Mougins
  - Centre Antoine Lacassagne, Nice
  - Hopital Saint Louis, Paris
  - Hôpital Pitie Salpetriere, Paris
  - Chu Lyon Sud, Pierre-Bénite
  - INSTITUT de CANCEROLOGIE DE L'OUEST - site René Gauducheau, Saint-Herblain
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared at an individual level. Those data will be part of the study database including all enrolled patients.